CLINICAL TRIAL: NCT04101903
Title: Evaluation of Aid to Diagnosis for Congenital Dysplasia of the Hip in General Practice: Controlled Randomised Trial
Brief Title: Evaluation of Aid to Diagnosis for Congenital Dysplasia of the Hip in General Practice
Acronym: HipDyS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: University College, London (Other); University of Bedfordshire (Other); King's College London (Other); Steps Charity Worldwide (Unknown); Longrove Surgery (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 19IR05; RP-PG-0616-20006 (Other: Great Ormond Street Hospital NHS Foundation Trust)
Record Dates: First submitted 2019-09-17; First posted 2019-09-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Developmental Dysplasia of the Hip
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diagnostic Aid (Experimental): The experimental group will use the trial diagnostic aid for all 6-week infant hip checks
  Interventions: Diagnostic Test: The 6-week Hip Checklist
- Standard of Care (No Intervention): The control group will assess infants according to standard practice, during the 6-week hip check.

INTERVENTIONS:
Diagnostic Test: The 6-week Hip Checklist — Comprehensive 9-item structured guide to aid in correct diagnosis of developmental dysplasia of the hip.
  Arms: Diagnostic Aid

SUMMARY:
Developmental dysplasia of the hip (DDH) is one of the most common inborn diseases. Early diagnosis of this condition is very important and it can be harmful both to miss DDH and label normal infants as having DDH. Why DDH can be missed or labelled to normal children is not well understood but can be related to the doctor's knowledge, skill and the way the hip consultation is conducted. This research aims to help overcome these issues and proposes the use of a diagnostic aid (checklist) for DDH in general practices (GP).

The Investigator will divide general practices (GP) in England into two groups. One group will use our checklist for all hip checks they carry out. The other group will work as they usually do, without the aid. The study wishes to compare if GPs who use the checklist will do better in identifying babies with DDH than those who do not use our checklist. The Investigator will also evaluate whether using the checklist reduces costs for families around trips to doctors or hospitals, and costs to the NHS (National Health Service). In addition The Investigators will interview general practitioners, health visitors and carers of infants to elicit their perceptions about the intervention.

The study will include GPs registered in England who carry out the 6-week hip check and agree to being randomised and to hospitals releasing data on infants they had examined during the study period. Practices planning to close within 12 months of the start of the study are not eligible. Eligible infants will be identified by general practice patient registers and infants will be invited to attend a 6-week check at their local practices, the research sites. The study plans to include a total of 152 practices in this study and will collaborate with 15 NIHR (National Institute of Health Research) CRNs (Clinical Research Network) to recruit GP practices with efficient and existing infrastructure.

DETAILED DESCRIPTION:
1. Objectives:

   * To determine whether the use of a check list for the 6-week hip check can (i) reduce the number of clinically insignificant referrals from primary to secondary care, and (ii) reduce the number of Developmental dysplasia of the hip (DDH) diagnosed beyond the age of 12 weeks.
   * To determine the cost-effectiveness of this intervention considering a life time horizon.
   * To conduct an integrated qualitative and quantitative process evaluation in order to: understand the participants' experience with the intervention; identify how the intervention affects general practitioners' capability, opportunity and motivation in relation to the 6-week check; study how the intervention is implemented; and investigate how contextual factors affect uptake of the intervention.
2. Type of trial: Phase III, cluster randomised controlled trial
3. Trial design and methods: This trial incorporates (i) 4-months internal pilot in order to confirm realistic recruitment targets; (ii) process evaluation encompassing qualitative research on changing physician referral behaviour and on normalising the intervention in practice; and (iii) health economic evaluation.
4. Trial duration per participant: 24 months
5. Planned trial sites: 172 GP practices in England. Half will be randomised to the experimental arm (using the diagnostic aid) and half to the control arm (standard of care 6 week hip check)
6. Total number of participants planned: 172 GP practices will be randomised (with an average of 110 infants recruited across the trial period per practice).
7. Main inclusion criteria:

   * Inclusion: GP practices registered in England and who carry out the 6-week hip check as part of their routine work - these practices must be using either EMIS or System One clinical computer systems

ELIGIBILITY:
Inclusion Criteria:

* General practices (GP) registered in England and who carry out the 6-week infant hip check as part of their routine work.
* Practice using either EMIS or SystemOne clinical computer systems
* General practitioners recording all 6 week baby hip examination on their computer template
* GPs willing to give informed consent to (a) being randomized, (b) willing to undergo observations, interviews and questionnaires and (c)collaborating secondary care facilities releasing data about all infants undergoing the 6-week hip check GP practices during the duration of the randomised controlled trial.
* GPs conducting the 6 week check must agree to view the training video on the examination of babies' hips at 6 weeks at baseline
* In the study practice, infants who are eligible for this study will be those presenting to any of the practices if aged <11 weeks when the 6-week check is done in the GP practice.

Exclusion Criteria:

* Any GP practice that is to close down within 12 months of when the first patient would be recruited in this practice.
* Parents/carers aged under 18

Ages: 6 Weeks to 11 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Clinical Importance of referrals | 2 weeks following hip check
  Number of referred hips that are considered clinically insignificant (referrals resulting in reassurance and discharge from secondary care).

SECONDARY OUTCOMES:
Number of appropriate referrals per GP practice | Within 2 years of hip check
  Number of referred infants with a hip deemed clinically significant (any hip of an infant that warrants treatment, evaluation and/or monitored by secondary care specialist.
Number of Late diagnoses | Within 2 years of hip check
  Cases of developmental dysplasia of the hip that is diagnosed by a specialist secondary care facility at age 3-24 months.
Consequences of Late diagnoses | Within 2 years of hip check
  How the late diagnoses of developmental dysplasia of the hip affects the patients treatment. For example, whether they need more treatment than if it were to be detected early.
Volume of referrals | Within 2 years of hip check
  Total number of patients referred to secondary care in trial period
Timeliness of referrals | Within 2 years of hip check
  Number of days from general practitioner referral to consultation with orthopaedic specialist
Incremental costs of using aid | Within 2 years of hip check
  Costs associated with using aid per clinically insignificant referral avoided, per late diagnosis avoided, per quality of life in years gained and the net monetary benefit of using the tool.
Incidence of developmental dysplasia of the hip | Within 2 years of hip check
  Clinically significant cases of developmental hip dysplasia in the entire study period (any hip of an infant that warrants treatment, evaluation and/or monitored by specialist secondary care facility.
Impact of the intervention on general practitioner behaviour | Within 2 years of hip check
  GP behaviour in relation to 6-week hip check to be measured based on 14 domains of the adapted theoretical domains framework questionnaire. The 14 domains include knowledge, skills, social/professional role and identity, beliefs about capabilities, optimism, beliefs about consequences, reinforcement, intentions, goals, memory/attention and decision processes, environmental context and resources, social influences, emotion and behavioural regulation. Per domain the scale ranges from 1-10 of scoring (with 1 being the lowest and 10 the highest of agreement with the statements indicated).
Parent/Carer general worry at present | Within 2 weeks of hip check
  As measured by Spielberger State-Trait Anxiety Inventory 6-items short form. This comprises of 6 statements to be answered on a scale of 1 to 4 with 4 being the highest measure of anxiety.
Parent/Carer worry related to developmental dysplasia of the hip | Within 2 weeks of hip check
  As measured by Infant Hip Worries Inventory. This comprises of 12 statements to be answered on a scale of 1 to 5, with 1 being the lowest and 5 the highest.
Parent/Carer satisfaction with the trial intervention | Within 2 weeks of hip check
  As measured by EUROPEP Dimensions of care subscale. This comprises of 23 statements to be answered on a scale of 1 to 5, with 1 being the lowest possible rating and 5 the highest.
Parent/Carer acceptability of trial intervention | Within 2 weeks of hip check
  As measured by qualitative interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Rise Group Practice, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be used for publication.

REFERENCES:
- [Derived] Roposch A, Warsame K, Chater A, Green J, Hunter R, Wood J, Freemantle N, Nazareth I. Study protocol for evaluation of aid to diagnosis for developmental dysplasia of the hip in general practice: controlled trial randomised by practice. BMJ Open. 2020 Dec 2;10(12):e041837. doi: 10.1136/bmjopen-2020-041837. PMID 33268429